CLINICAL TRIAL: NCT06550310
Title: Nutrition and Body Composition and Association With Clinical Outcomes in Inflammatory Bowel Disease
Brief Title: Nutrition and Clinical Outcomes in IBD
Status: Not yet recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 337108
Record Dates: First submitted 2024-07-31; First posted 2024-08-13 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Malnutrition; Sarcopenia
Keywords: Body composition; Nutritional status; Nutritional markers; Nutritional screening tools; Nutritional assessment; Sarcopenia; Radiological muscle mass; Inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Malnutrition; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical treatment group: Patients with inflammatory bowel disease (Crohn's disease, ulcerative colitis or IBD-U) starting a new advanced medical therapy (e.g. biologic or small molecule)
- Surgical treatment group: Patients with inflammatory bowel disease (Crohn's disease, ulcerative colitis or IBD-U) undergoing an IBD-related surgery

SUMMARY:
The goal of this observational study is to demonstrate that nutritional status and body composition have an impact on clinical outcomes in inflammatory bowel disease (IBD).

The main objectives are:

1. To compare the detection rates of undernutrition between a range of nutritional screening tools, physiological measures and assessment tools amongst patients with different IBD phenotypes
2. To correlate nutritional status, nutritional biomarkers and body composition with clinical outcomes in patients with IBD treated with advanced medical therapy or surgery
3. To determine a potential relationship between radiological muscle mass measurements and clinical outcomes in patients with IBD treated with advanced medical therapy or surgery

Participants will undergo an assessment at pre-treatment baseline and then again at their scheduled follow-up. This is a non-interventional study and participants will not be required to have any invasive tests or hospital visits beyond that of standard clinical care.

DETAILED DESCRIPTION:
Background and Rationale:

Inflammatory bowel disease (IBD) comprises Crohn's disease (CD) and ulcerative colitis (UC). It affects nearly 400,000 people in the United Kingdom (UK) and the global prevalence is rising. Many patients suffer an impaired quality of life. Whilst advanced medical therapies are being used more often, the lifetime risk of surgery is as high as 70%. Unfortunately, loss of response to medical therapies and post-operative complications remain major clinical challenges. Risk factors for adverse treatment outcomes include disease duration, emergency surgery and undernutrition. Not only is undernutrition a risk factor for adverse clinical outcomes, it is present in up to 36% of patients with IBD. Crucially, unlike other risk factors, it is also modifiable with cheap and safe interventions. It therefore presents an ideal opportunity for intervention. Despite this, current methods of detecting undernutrition in IBD are unfit for purpose.

Body composition (BC) analysis is emerging as a highly clinically relevant physiological marker in IBD. Skeletal muscle loss with functional impairment (sarcopenia) in IBD patients is associated with a range of outcomes including disease flares, hospitalisation, need for surgery and need for ICU admissions. Radiological measurement of skeletal muscle index (SMI) at the level of the 3rd lumbar vertebra is objective and reproducible. Validated software designed specifically for this purpose (Slice-o-Matic [Tomovision, Canada]) can be used on CT/MRI scans which are often performed as part of standard IBD care. However, despite this, BC analysis by any method is not performed in routine clinical practice. The most commonly used physiological markers in the UK remain weight and body mass index (BMI), which do not provide any measure of BC.

Overall, there remains uncertainty over which nutritional tools should be used in patients with IBD. Most studies have been small, retrospective and heterogenous. No study has performed a comparative analysis of more than three measurements in the same patient cohort. Evidence of the ability of widely used nutritional screening tools to identify IBD patients most at risk of adverse clinical outcomes is lacking. Finally, there is little data describing the performance of different tools and measures according to disease phenotype and disease activity. This study proposes to meet this knowledge gap by comparing a range of nutritional tools in a large, prospective, well-phenotyped IBD cohort.

Study design:

Eligible patients will be identified from dedicated IBD multi-disciplinary weekly meetings, IBD clinic, medical infusion suites and the medical records. The clinical team will be aware of the study and can also flag potential eligible patients to the investigators. Participants will be contacted or approached directly in clinic or via telephone.

This will be a prospective, non-interventional study performed at Barts Health National Health Service (NHS) Trust over 4 years. For patients treated with advanced medical therapies, the entire prospective dataset will be collected at a pre-treatment baseline (within 4 weeks before treatment) and at weeks 14 and 52 after therapy commencement. For patients undergoing surgery, data will be collected at a pre-operative baseline (within 4 weeks before surgery) and at 3 months post-operatively. Data relating to dietetic input and artificial nutritional support will be included. The following outcomes from medical therapy will be collected at weeks 14 and 52: clinical response, clinical and biochemical remission, corticosteroid use, therapy switch, IBD-surgery. The following surgical outcomes will be collected: length of post-operative stay, formation of unplanned stoma, 30-day complication rate, 30-day complication grade (defined by the Clavien-Dindo scale) and 90-day readmission rate. Participants will then be followed-up longitudinally over the aforementioned defined timepoints. Muscle mass measurements will be performed by exporting CT/MRI image slices at the level of the third vertebra from Trust computers and using Slice-O-Matic software to measure skeletal muscle indices (SMI). Additionally, we will access de-identified CT/MRI scans from 946 well-phenotyped patients who have undergone IBD surgery collected by the national UK IBD Bioresource and made available via the Gut Reaction initiative hosted by the National Institute for Health and Care Research (NIHR). Post-operative outcome data will also be available, enabling this to be used as an external validation cohort to the primary surgical dataset. Within the internal cohort, handgrip strength and timed up and go test (TUG) or gait speed will be performed prospectively at scheduled visits, to assess muscle strength and physical performance respectively. All nutritional parameters collected will be correlated with clinical outcomes.

The clinical data that will be collected is outlined below:

Demographics: age, gender, ethnicity, comorbidities, smoking status, postcode IBD phenotype: diagnosis, duration, disease location and behaviour (CD), disease extent (UC) IBD treatment: current IBD therapy (>3 months), previous IBD therapy, previous IBD-related surgery IBD activity: Harvey Bradshaw Index (HBI) or partial Mayo scores, C-reactive protein (CRP), faecal calprotectin Nutritional screening tools: Malnutrition Universal Screening Tool (MUST), Nutrition Risk Screening Tool-2002 (NRS-2002), Malnutrition Inflammation Risk Tool (MIRT) Nutritional assessment tools: Subjective Global Assessment (SGA), Global Leadership Initiative on Malnutrition (GLIM) criteria Weight, height, BMI, anthropometry (waist circumference, mid-upper arm circumference, triceps skinfold thickness, mid-arm muscle circumference) Handgrip strength Timed up and go test (TUG) or gait speed Bioelectrical impedance analysis, including skeletal muscle mass (kg), body fat (%) and visceral adiposity (kg) Blood tests: Haemoglobin, folate, ferritin, B12, vitamin D, zinc, copper, selenium Dietetics: dietetic review, special diets, presence and type of artificial nutritional support Food intake (24-hour food diaries) Food frequency questionnaire Food-related quality of life questionnaire Skeletal muscle index

The end of recruitment will be month 18 for the medical arm and month 27 for the surgical arm, to allow sufficient time for follow-up and data analysis. The End of Study will be defined as the conclusion of follow-up monitoring, data analysis and write-up at month 36.

Analysis:

Descriptive statistics will be taken at baseline for both medical and surgical cohorts. These exploratory variables will be measured at the three timepoints (as outlined above) to compare if any statistically significant difference is present. Statistical significance will be considered if a threshold of p=0.05. One-way repeated measures analysis of variance (ANOVA) will be performed for both groups.

Further sub-group analysis to determine correlations between the exploratory variables and outcomes will be performed using multi-linear and binary logistic regression. Standard demographical analysis will be collected and further sub-group analysis based on ethnicity may be performed.

Ethical approval has been obtained from the Health Research Authority.

This study is sponsored by Barts Health NHS Trust.

There are no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease (Crohn's disease, ulcerative colitis or IBD-U) starting a new advanced medical therapy
* Patients with inflammatory bowel disease (Crohn's disease, ulcerative colitis or IBD-U) undergoing an IBD-related surgery
* Age >16
* Patients able and willing to provide written informed consent

Exclusion Criteria:

* Patients below the age of 16
* Patients who cannot provide informed consent
* Patients with a cardiac pacemaker or internal defibrillator
* Patients with active cancer and other disorders associated with severe cachexia

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults (>16) with a diagnosis of inflammatory bowel disease (IBD) attending a tertiary IBD centre who are undergoing a new treatment or change in treatment, or an operation for their condition
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of nutritional parameters (at baseline and during treatment) with pre-defined clinical outcomes in patients undergoing advanced medical therapy (at 14 and 52 weeks). | 14 and 52 weeks
  Clinical outcomes are as follows clinical response, clinical and biochemical remission, corticosteroid use, therapy switch or IBD related-surgery.
  Clinical response in UC is defined as a ≥2-point and ≥30% decrease from baseline in partial Mayo score and a ≥1-point decrease from baseline in rectal bleeding sub-score or an absolute rectal bleeding sub-score ≤1. Clinical response in CD is defined as ≥ 3 points decrease of HBI score. Clinical remission is defined as a partial Mayo score of 0-1 in UC or HBI of ≤4 in CD. Biochemical remission is defined as faecal calprotectin <200μg/mg and CRP ≤5mg/L.
Correlation of nutritional parameters (at baseline and during treatment) with pre-defined clinical outcomes in patients undergoing IBD-related surgery (at 30 and 90 days). | 30 and 90 days
  Clinical outcomes are defined as length of post-operative stay, formation of unplanned stoma, 30-day complication rate, 30-day complication grade (defined by the Clavien-Dindo scale) and 90-day readmission rate.

SECONDARY OUTCOMES:
Correlation of currently used radiological muscle mass thresholds with pre-defined clinical outcomes in patients undergoing advanced medical therapy (at 14 and 52 weeks). | 14 and 52 weeks
  Clinical outcomes are as follows clinical response, clinical and biochemical remission, corticosteroid use, therapy switch or IBD related-surgery.
  Clinical response in UC is defined as a ≥2-point and ≥30% decrease from baseline in partial Mayo score and a ≥1-point decrease from baseline in rectal bleeding sub-score or an absolute rectal bleeding sub-score ≤1. Clinical response in CD is defined as ≥ 3 points decrease of HBI score. Clinical remission is defined as a partial Mayo score of 0-1 in UC or HBI of ≤4 in CD. Biochemical remission is defined as faecal calprotectin <200μg/mg and CRP ≤5mg/L.
Correlation of currently used radiological muscle mass thresholds with pre-defined clinical outcomes in patients undergoing advanced IBD-related surgery (at 30 and 90 days). | 30 and 90 days
  Clinical outcomes are defined as length of post-operative stay, formation of unplanned stoma, 30-day complication rate, 30-day complication grade (defined by the Clavien-Dindo scale) and 90-day readmission rate.

CONTACTS AND LOCATIONS:
Overall Officials: Shameer Mehta, MD, Principal Investigator — Barts & The London NHS Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Inflammatory Bowel Disease Collaborators. The global, regional, and national burden of inflammatory bowel disease in 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Gastroenterol Hepatol. 2020 Jan;5(1):17-30. doi: 10.1016/S2468-1253(19)30333-4. Epub 2019 Oct 21. PMID 31648971
- [Background] Knowles SR, Graff LA, Wilding H, Hewitt C, Keefer L, Mikocka-Walus A. Quality of Life in Inflammatory Bowel Disease: A Systematic Review and Meta-analyses-Part I. Inflamm Bowel Dis. 2018 Mar 19;24(4):742-751. doi: 10.1093/ibd/izx100. PMID 29562277
- [Background] Lewis RT, Maron DJ. Efficacy and complications of surgery for Crohn's disease. Gastroenterol Hepatol (N Y). 2010 Sep;6(9):587-96. PMID 21088749
- [Background] Gklavas A, Dellaportas D, Papaconstantinou I. Risk factors for postoperative recurrence of Crohn's disease with emphasis on surgical predictors. Ann Gastroenterol. 2017;30(6):598-612. doi: 10.20524/aog.2017.0195. Epub 2017 Sep 26. PMID 29118554
- [Background] Ma C, Moran GW, Benchimol EI, Targownik LE, Heitman SJ, Hubbard JN, Seow CH, Novak KL, Ghosh S, Panaccione R, Kaplan GG. Surgical Rates for Crohn's Disease are Decreasing: A Population-Based Time Trend Analysis and Validation Study. Am J Gastroenterol. 2017 Dec;112(12):1840-1848. doi: 10.1038/ajg.2017.394. Epub 2017 Oct 31. PMID 29087396
- [Background] Ananthakrishnan AN, Shi HY, Tang W, Law CC, Sung JJ, Chan FK, Ng SC. Systematic Review and Meta-analysis: Phenotype and Clinical Outcomes of Older-onset Inflammatory Bowel Disease. J Crohns Colitis. 2016 Oct;10(10):1224-36. doi: 10.1093/ecco-jcc/jjw054. Epub 2016 Feb 29. PMID 26928965
- [Background] Nguyen GC, Munsell M, Harris ML. Nationwide prevalence and prognostic significance of clinically diagnosable protein-calorie malnutrition in hospitalized inflammatory bowel disease patients. Inflamm Bowel Dis. 2008 Aug;14(8):1105-11. doi: 10.1002/ibd.20429. PMID 18302272
- [Background] Ananthakrishnan AN, McGinley EL, Binion DG, Saeian K. A novel risk score to stratify severity of Crohn's disease hospitalizations. Am J Gastroenterol. 2010 Aug;105(8):1799-807. doi: 10.1038/ajg.2010.105. Epub 2010 Mar 9. PMID 20216534
- [Background] Ciocirlan M, Ciocirlan M, Iacob R, Tantau A, Gheorghe L, Gheorghe C, Dobru D, Constantinescu G, Cijevschi C, Trifan A, Goldis A, Diculescu M. Malnutrition Prevalence in Newly Diagnosed Patients with Inflammatory Bowel Disease - Data from the National Romanian Database. J Gastrointestin Liver Dis. 2019 Jun 1;28:163-168. doi: 10.15403/jgld-176. PMID 31204412
- [Background] Casanova MJ, Chaparro M, Molina B, Merino O, Batanero R, Duenas-Sadornil C, Robledo P, Garcia-Albert AM, Gomez-Sanchez MB, Calvet X, Trallero MDR, Montoro M, Vazquez I, Charro M, Barragan A, Martinez-Cerezo F, Megias-Rangil I, Huguet JM, Marti-Bonmati E, Calvo M, Campdera M, Munoz-Vicente M, Merchante A, Avila AD, Serrano-Aguayo P, De Francisco R, Hervias D, Bujanda L, Rodriguez GE, Castro-Laria L, Barreiro-de Acosta M, Van Domselaar M, Ramirez de la Piscina P, Santos-Fernandez J, Algaba A, Torra S, Pozzati L, Lopez-Serrano P, Arribas MDR, Rincon ML, Pelaez AC, Castro E, Garcia-Herola A, Santander C, Hernandez-Alonso M, Martin-Noguerol E, Gomez-Lozano M, Monedero T, Villoria A, Figuerola A, Castano-Garcia A, Banales JM, Diaz-Hernandez L, Arguelles-Arias F, Lopez-Diaz J, Perez-Martinez I, Garcia-Talavera N, Nuevo-Siguairo OK, Riestra S, Gisbert JP. Prevalence of Malnutrition and Nutritional Characteristics of Patients With Inflammatory Bowel Disease. J Crohns Colitis. 2017 Dec 4;11(12):1430-1439. doi: 10.1093/ecco-jcc/jjx102. PMID 28981652
- [Background] Bamba S, Sasaki M, Takaoka A, Takahashi K, Imaeda H, Nishida A, Inatomi O, Sugimoto M, Andoh A. Sarcopenia is a predictive factor for intestinal resection in admitted patients with Crohn's disease. PLoS One. 2017 Jun 23;12(6):e0180036. doi: 10.1371/journal.pone.0180036. eCollection 2017. PMID 28644887
- [Background] Zhang T, Cao L, Cao T, Yang J, Gong J, Zhu W, Li N, Li J. Prevalence of Sarcopenia and Its Impact on Postoperative Outcome in Patients With Crohn's Disease Undergoing Bowel Resection. JPEN J Parenter Enteral Nutr. 2017 May;41(4):592-600. doi: 10.1177/0148607115612054. Epub 2015 Oct 15. PMID 26471990
- [Background] Pedersen M, Cromwell J, Nau P. Sarcopenia is a Predictor of Surgical Morbidity in Inflammatory Bowel Disease. Inflamm Bowel Dis. 2017 Oct;23(10):1867-1872. doi: 10.1097/MIB.0000000000001166. PMID 28604415
- [Background] Peng P, Hyder O, Firoozmand A, Kneuertz P, Schulick RD, Huang D, Makary M, Hirose K, Edil B, Choti MA, Herman J, Cameron JL, Wolfgang CL, Pawlik TM. Impact of sarcopenia on outcomes following resection of pancreatic adenocarcinoma. J Gastrointest Surg. 2012 Aug;16(8):1478-86. doi: 10.1007/s11605-012-1923-5. Epub 2012 Jun 13. PMID 22692586
- [Background] Lomer MC, Gourgey R, Whelan K. Current practice in relation to nutritional assessment and dietary management of enteral nutrition in adults with Crohn's disease. J Hum Nutr Diet. 2014 Apr;27 Suppl 2:28-35. doi: 10.1111/jhn.12133. Epub 2013 Jun 13. PMID 23763616